CLINICAL TRIAL: NCT02809092
Title: A Phase I/II Clinical Trial Testing the Safety and Feasibility of IL-21- Expanded Natural Killer Cells for the Induction of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Interleukin-21 (IL-21)- Expanded Natural Killer Cells for Induction of Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0457
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia, Natural Killer Cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — IL32 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK Cells + Chemotherapy Starting (Experimental): Starting on Day -7, G-CSF daily by vein until post nadir of absolute neutrophil counts (ANC) are equal or over 1000. Day -6 to Day -2 Fludarabine administrated by vein at 30 mg/m^2. Four hours later Cytarabine administrated by vein at 2 g/m^2. Natural killer (NK) cell infusion Days 0 to 14 for 6 doses total. The first group of participants receive lowest dose level. Each new group receives a higher dose than the group before it, if no intolerable side effects were seen. This will continue for up to 6 dose levels or until the highest tolerable dose of NK cells is found. One (1) to 10 participants will be treated in each dose level.
  NK Cell infusion on Days 0 to 14 for 6 doses total according to dose escalation schema.
  Interventions: Biological: NK Cells + Chemotherapy Starting

INTERVENTIONS:
Biological: NK Cells + Chemotherapy Starting — Drug: G-CSF G-CSF daily by vein starting on Day -7 until post nadir of absolute neutrophil counts (ANC) are equal or over 1000.
  Other Names:
  Filgrastim Neupogen Drug: Fludarabine monophosphate 30 mg/m2 by vein on Days -6, -5, -4, -3, and -2.
  Other Names:
  Fludarabine Phosphate Fludara Drug: Cytarabine 2 g/m^2 by vein on Days -6, -5, -4, -3, and -2.
  Other Names:
  Ara-C Cytosar DepoCyt Cytosine arabinosine hydrochloride Procedure: Natural Killer (NK) Cell Infusion NK Cell infusion on Days 0 to 14 for 6 doses total according to dose escalation schema.
  Other Names: Natural killer cells

SUMMARY:
Relapsed acute myeloblastic leukemia (AML) requires remission prior to allogeneic Hematopoietic Stem Cell Transplant (HSCT) for optimal survival, but is a disease with poor response to chemotherapy. Human leukocyte antigen (HLA) haploidentical, Natural killer (NK) enriched peripheral blood cell infusions have shown safety in patients with poor prognosis AML. Though not powered for such an assessment, this trial showed a promising but not statistically significant trend in remission rate. NK cell therapy was limited by small numbers of NK cells attainable through leukapheresis. We have now demonstrated that large numbers of NK cells can be propagated ex vivo from a small volume blood draw, obviating the need for donor leukapheresis. The purpose of this trial is to determine the feasibility and maximum tolerated dose of expanded NK cells and estimate the toxicity of treating relapsed/refractory AML with fludarabine + high-dose cytarabine + G-CSF (FLAG) chemotherapy followed by haploidentical expanded natural killer (NK) cells.

The first NK cell dosing cohort will be well below the currently-established safe dose of pheresis-derived NK cells, as expanded NK cells may have increased toxicity because of their activated phenotype. In order to avoid accruing patients at suboptimal doses, a dose escalation schema based on the principles of an accelerated titration design is used in this study to allow expeditious advancement up to the current safe dose of NK cells.

DETAILED DESCRIPTION:
While growing the NK cells from the blood in the lab, mismatched T cells may also grow, which can cause a reaction against normal tissue called graft-vs-host disease (GvHD). In the lab, the T cells will be removed from the cell product using special magnets and antibody-coated magnetic beads. The drug aldesleukin (interleukin-2) is then added to the NK cells to improve their function. The aldesleukin will be washed out of the cell product before it is given to you.

The NK cells will be donated from a family member who has a certain genetic type in their blood called HLA that partly matches yours.

If you agree to take part in this study, you will be assigned to a dose level of NK cells based on when you joined this study. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue for up to 6 dose levels or until the highest tolerable dose of NK cells is found. One (1) to 10 participants will be treated in each dose level.

The day you receive the first NK cell infusion is called Day 0. The days before you receive your NK cell infusion are called minus days (D-). The days after you receive the NK cell infusion are called plus days (D+).

Study Drug Administration:

On Day -7, you will be admitted to the hospital and given fluids by vein to hydrate you.

On Days -6, -5, -4, -3, and -2, you will receive fludarabine by vein over about 30 minutes. About 4 hours later, you will receive cytarabine by vein over about 1 hour. If you are 60 years old or older, you will "rest" (not receive chemotherapy) on Day -2.

On Day -1, you will rest.

Three (3) times a week for 2 weeks, you will receive NK cells by vein over 30 minutes. You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

You will receive filgrastim as an injection under the skin 1 time a day, starting on Day -7 and continuing until your white blood cell levels are high enough. Filgrastim is designed to help with the growth of white blood cells.

Study Visits:

Before treatment starts:

Your medical history will be recorded. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).

Blood (about 2 teaspoons) will be drawn for routine tests.

Before each NK cell infusion:

Your medical history will be recorded. You will have a physical exam, including measurement of your vital signs. Blood (about 2 teaspoons) will be drawn for routine tests. The amount of oxygen in your blood will be measured by placing a sensor on the tip of your finger.

Twice a week, while your blood counts are low, you will have blood (about 2 teaspoons) drawn for routine tests.

Once your blood counts are high enough, you will have blood (about 2 teaspoons) drawn for routine tests once a week until Day +56.

Once your blood counts are high enough or around Day +28 (whichever is earlier), you will have a bone marrow aspiration and biopsy to check the status of the disease and DNA tests to check if the cells in your bone marrow are yours or your NK cell donor's. To collect a bone marrow aspiration/biopsy, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

Blood (about 2 teaspoons) will be drawn to test the genetic makeup and function of the infused NK cells and to check the status of the disease:

Before treatment starts. Before and about 1-3 hours after each NK cell infusion. Once a day on Days +14, +16, +18, +21, and then weekly until Day +56.

Length of Study:

Your participation on the study will be over on Day +56.

You will be taken off study early if the disease gets worse, if intolerable side effects occur, if not enough NK cells can be collected, or if you are unable to follow study directions.

This is an investigational study. Cytarabine, fludarabine, and filgrastim are FDA approved and commercially available for the treatment of AML. The investigational part of this study is to find the best dose of NK cells that can be given with the goal of helping to prevent the cancer from coming back. The way the researchers process the NK cells is investigational and is not FDA approved.

Up to 30 patients will take part in this study. All will be enrolled at Cellular Therapy Center (HCPA)

ELIGIBILITY:
Inclusion Criteria:

Obtained within 30 days prior to beginning the lymphodepleting conditioning regimen, unless otherwise specified.

* Patients with relapsed AML, including Canadian Neurological Scale (CNS) disease or previous hematopoietic stem cell transplantation, which has failed remission to at least one cycle of standard or experimental reinduction chemotherapy, or primary refractory AML (primary AML that has failed remission to at least two cycles of induction therapy)
* Availability of a haploidentical family peripheral blood donor selected for best possible killer cell inhibitory receptor (KIR) reactivity.
* Patient age between 2 and 59 years, inclusive.
* Patient must have recovered from the treatment-related toxicities of prior cytotoxic agents received in the 4 weeks prior to beginning treatment on this protocol, with the exception of cytopenias resulting from persistent disease, and alopecia.
* "Zubrod" performance scale ≤ 2 or "Lansky" scale ≥ 60.
* Adequate renal function defined as:

  * Serum creatinine ≤2 mg/dL for adults.
  * Serum creatinine ≤2 mg/dL or ≤2 times upper limit of normal (ULN) for age (whichever is less) for children.
  * Or, if serum creatinine does not meet above criteria, patient will be eligible if 24h creatinine clearance ≥60 mL/min/1.73m2.
* Adequate liver function, defined as: Total bilirubin ≤2 mg/dL and serum glutamate pyruvate transaminase(SGPT) (ALT) ≤2.5 x ULN for age (unless Gilbert's disease or abnormal liver function due to primary disease).
* Pulmonary symptoms controlled by medication and pulse oximetry ≥ 92% room air.
* New York Heart Association classification < III
* Negative serum test to rule out pregnancy within 2 weeks prior to registration in females of childbearing potential (non childbearing potential defined as premenarchal, greater than one year post-menopausal, or surgically sterilized).
* Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator.
* Negative serology for human immunodeficiency virus (HIV).

Exclusion Criteria:

* Failed attaining remission with any previous FLAG therapy.
* Investigational therapies in the 4 weeks prior to beginning treatment on this protocol.
* Congestive heart failure <6 months prior to screening
* Unstable angina pectoris <6 months prior to screening
* Myocardial infarction <6 months prior to screening

Ages: 2 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of membrane-bound interleukin 21 (mbIL21)-Expanded Haploidentical NK Cells After Induction Chemotherapy with Fludarabine, Cytarabine, and Granulocyte-colony stimulating factor (G-CSF). | 28 days
  Maximum tolerated dose defined as highest dose studied in which 6 patients have been treated and at most 2 patients with dose-limiting toxicities (DLTs) observed.
  A dose-limiting toxicity (DLT) is defined as:
  Acute severe (grade 3 or 4) infusional allergic reaction related to the NK cells infusion.
  Prolonged cytopenia beyond D+28. If neutropenia is still present at day 28, that will trigger the designation of prolonged neutropenia as a DLT. If neutrophil counts have recovered by day 28, then no DLT will have occurred. In either case, the status of neutrophil recovery beyond day 28 will not change the designation of DLT or No DLT made at day 28.
  Acute GvHD overall grade 3 or 4. Severe (grade 3 or 4) unexpected toxicity related to the NK cell infusion.

SECONDARY OUTCOMES:
Complete Remission (CR) Assessment Following Infusion of the NK Cells | Baseline up to Day 56
  Percentage of participants with complete remission (CR): Bone marrow aspiration - Less than 5% leukemic blasts. Disease assessment after neutrophil recovery and or Day 28, whichever is earlier: 1. Unilateral bone marrow biopsy and aspirate for cytology, flow cytometry, Minimal Residual Disease MRD, chimerism, cytogenetics, and fluorescent in situ hybridization (FISH) (for known tumor markers). 2. If recovery has not occurred by Day +28, then a second bone marrow will be obtained at the time of neutrophil recovery or Day +56, whichever is earlier. CR estimated with Kaplan-Meier estimator and tabulated with 95% confidence intervals.
Donor NK-Cell Expansion | 28 days
  Donor NK-cell expansion defined as an absolute circulating donor-derived NK cell count that increases above the post-infusion level. Proportion of patients with successful in vivo NK-cell expansion estimated with a 95% confidence interval. The following chimerism methods employed to determine origin and number of circulating NK cells. Chimerism may be determined by flow cytometry using haplotype-specific antibodies. Chimerism may be determined by short tandem repeat (STR) polymorphisms. When there is a sex-mismatch between the donor and the recipient, assays based on determining the frequency of sex-chromosomes may be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Silla, Doctor, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Centro Terapia e Tecnologia Celular, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided